CLINICAL TRIAL: NCT05106543
Title: Immediate Effect Of Kinesiological Taping On Functionality In Hemiplegic Patients
Brief Title: Immediate Effect Of Kinesiological Taping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, mustafa gulsen, assocc.prof., Baskent University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BaskentU 1
Record Dates: First submitted 2021-10-12; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Hemiplegia
Keywords: Hemiplegia; Kinesiology taping; Functionality
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesiologic tape (Experimental): first group of 20 people (experimental group) T max branded kinesiology tape was applied to both M. Quadriceps Femoris and M. Gastrocnemius muscles of the experimental group.
  Timed get up and go test was applied to evaluate functionality. All evaluations were applied before taping, immediately after taping and 45 minutes after taping. Patients in both groups were asked not to have their tapes removed until the 4th day. Apart from routine physical therapy methods and taping, no other treatment was applied to the patients.
  Interventions: Device: Immediate Effect Of Kinesiological Taping On Functionality In Hemiplegic Patients
- patch tape (Placebo Comparator): second group of 20 people (control group) Roll branded patch tape was applied to both M. Quadriceps Femoris and M. Gastrocnemius muscles of the control group.
  Timed get up and go test was applied to evaluate functionality. All evaluations were applied to both groups before taping, immediately after taping and 45 minutes after taping. Patients in both groups were asked not to have their tapes removed until the 4th day. Apart from routine physical therapy methods and taping, no other treatment was applied to the patients.
  Interventions: Device: Immediate Effect Of Kinesiological Taping On Functionality In Hemiplegic Patients

INTERVENTIONS:
Device: Immediate Effect Of Kinesiological Taping On Functionality In Hemiplegic Patients — Kinesiological Taping

SUMMARY:
In this study, it is aimed to examine the immediate effect of kinesiological taping on functionality in hemiplegic patients. 40 hemiplegic patients with a mean age of 63±15 years were included to the study. The patients were divided into two groups using the computerized randomization method. Kinesiology tape was applied to the 1st group (study group), and a patch tape was applied to the 2nd group (control group). The demographic and physical characteristics of the people who agreed to participate in the study were recorded. In both groups; before taping, right after taping, 45 min. after and 4 days after taping Timed Get Up and Go Test (TUG) were administered. Both groups were asked not to remove the tapes at the end of the 4th day.

ELIGIBILITY:
Inclusion Criteria:

* agree to participate in the study after detailed information about the study,
* to have sufficient cognitive functions, to be diagnosed with hemiplegia by a specialist physician,
* to be 18 years of age or older

Exclusion Criteria:

* Diagnosis of other neurological diseases (Parkinson's, Multiple Sclerosis, etc.),
* cancer other than hemiplegia, heart failure, surgery in the area to be applied,
* vascular problems in the lower extremity,
* chronic kidney failure,
* infection.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Immadiate Effect Of Kinesiological Taping | 4 days
  With a computerized randomization system, 40 people, 20 of whom we applied kinesiology taping in the first group (study group), and the second group of 20 people (control group), were determined. T max branded kinesiology tape was applied to both M. Quadriceps Femoris and M. Gastrocnemius muscles of the experimental group. Roll branded plaster tape was applied to both M. Quadriceps Femoris and M. Gastrocnemius muscles of the control group.
  Timed get up and go test was applied to evaluate functionality. All evaluations were applied to both groups before taping, immediately after taping and 45 minutes after taping. Patients in both groups were asked not to have their tapes removed until the 4th day. All patients were re-evaluated on the 4th day. Apart from routine physical therapy methods and taping, no other treatment was applied to the patients.

CONTACTS AND LOCATIONS:
Overall Officials: emine atici, pt phd, Principal Investigator — Okan University
Locations (2):
- Turkey (Türkiye) (2):
  - Immediate Effect Of Kinesiological Taping On Functionality In Hemiplegic Patients, Istanbul
  - Okan University, Istanbul

IPD SHARING:
Plan to Share IPD: No